CLINICAL TRIAL: NCT06836804
Title: Validity and Reliability Study of the Turkish Long and Short Forms of the Cardiac Depression Scale
Brief Title: Validity and Reliability of the Turkish Version of the Cardiac Depression Scale
Acronym: TURK-CDS
Status: Enrolling by invitation | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Selcuk OZTURK, Associate Professor, MD, Kırıkkale University
Other Study IDs: 2025.01.11
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases; Depression
Keywords: Cardiovascular Diseases; Depression
MeSH Terms: conditions — Cardiovascular Diseases; Depression | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with CVDs: The study cohort includes participants with stable cardiovascular disease (CVD) condition who apply to outpatient cardiology clinics of Kırıkkale University Faculty of Medicine.
  Interventions: Other: Sociodemographic Data Form; Other: Short Form Health Survey; Other: Hospital Anxiety and Depression Scale; Other: Illness Intrusiveness Ratings Scale; Other: Cardiac Depression Scale

INTERVENTIONS:
Other: Sociodemographic Data Form — After inquiring about participants' sociodemographic characteristics, such as name, contact information, age, gender, marital status, education level, income, and place of residence, measurements of height, weight, and waist circumference will be obtained. Then, participants' CVD, psychiatric and other medical conditions, CVD risk factors, health history, and medications they are using will be queried. This information will be recorded in the sociodemographic data form. The sociodemographic data form has been prepared by the researchers.
Other: Short Form Health Survey — SF-36 is a self-assessment scale and can be completed in five minutes. SF-36 can evaluate both the negative and positive aspects of health. The scale consists of 36 items which are used to assess different health dimensions in 8 subscales: Physical functioning (10 items), social functioning (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items), and general health perception (5 items).
Other: Hospital Anxiety and Depression Scale — The HADS was designed in 1983 to identify anxiety and depression in individuals with physical illnesses. The HADS is a self-reported scale consisting of seven items each for the anxiety and depression subscales. Each item is scored from 0 to 3, and the total score for the anxiety and depression subscales is 21 points. The overall HADS score is obtained by summing the points from both subscales. A total subscale score between 0-7 indicates a normal test result, 8-10 indicates mild anxiety or depression, 11-15 indicates moderate anxiety or depression, and 16-21 indicates severe anxiety or depression. Higher scores represent higher levels of anxiety or depression, and the total HADS score reflects an overall measure of psychological distress. The survey can be completed in 2-5 minutes.
Other: Illness Intrusiveness Ratings Scale — The IIRS is an easy-to-administer scale designed to predict the psychosocial impact of chronic illness and to document and compare the effectiveness of therapeutic interventions. It consists of 13 questions which are completed by the patient. The scale measures how the limitations imposed by chronic and life-threatening diseases hinder participation in regular activities across 13 important aspects of life: Health, diet, work, active recreation (sports), passive recreation (reading, listening to music), finances, relationships with partners, sexual life, family relationships, other social relationships, self-expression/development, religious expression, and community and civic participation.
Other: Cardiac Depression Scale — CDS was designed to identify depression in individuals with CVDs. It consists of 26 items across 7 subscales. The subscales address issues such as sleep, uncertainty, mood, hopelessness, immobility, anhedonia, and cognition. The CDS is rated on a 7-point Likert scale, with seven items being reverse-coded. Based on patient feedback and clinical experience, two short forms were developed, each consisting of five questions. Both short forms showed good consistency with the original CDS. The first short form includes questions from the original CDS numbered 12, 24, 21, 10, and 9. The second short form includes questions from the original CDS numbered 12, 4, 25, 21, and 7.

SUMMARY:
The Cardiac Depression Scale (CDS) in both its long and short forms has been validated in various languages and populations and is used to detect depression in individuals with cardiovascular disease (CVD). However, there is no validity and reliability study of the CDS for CVD patients in the Turkish population available in the literature, which prevents its use in Turkish population. The study aims to test the validity and reliability of the Turkish version of long and short forms of the CDS in Turkish individuals with CVD.

DETAILED DESCRIPTION:
CVDs are among the leading causes of death worldwide and in Türkiye. Studies have shown that the prevalence of depression is higher among individuals with CVD compared to the general population. For example, higher rates of depression have been reported in patients who have undergone coronary bypass surgery, individuals who experienced myocardial infarction, and those with angina pectoris. Depression itself can be a cause of CVD, while CVD can also trigger depressive symptoms.

The presence of depression in individuals with CVD is associated with diverse adverse outcomes including mortality. Therefore, routine depression screening is recommended for individuals with CVD. Many scales are currently used in clinical practice for depression screening. The CDS was specifically developed in 1996 for individuals with CVD and remains the only scale in the literature designed for this purpose. The CDS consists of 26 self-administered items and is used to identify and assess the severity of depressive symptoms, including emotional, cognitive, and somatic characteristics. Originally developed in English in Australia, the scale has undergone validity and reliability studies for individuals with different CVD conditions across various languages and cultures. The CDS takes approximately five minutes to administer and score, and demonstrates robust psychometric properties in distinguishing mild, moderate, and severe depression. CDS scores range from 26 to 182 with higher scores indicating more severe depressive symptoms. A score of 95 or higher on the CDS can detect major depression in individuals with CVD with 85% specificity and 97% sensitivity.

Due to constraints such as time, resources, and personnel in clinical practice, two shorter forms of the CDS have been developed, each consisting of five items derived from the original scale. These short forms have also been validated in English for different CVD populations. However, no validity or reliability study of the CDS, in either its long or short forms, has been studied in Turkish population. Furthermore, the short forms of the CDS have not undergone validity and reliability analyses in any language other than English.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older and providing written consent to participate in the study
* Diagnosed with any cardiovascular disease (coronary artery disease, peripheral artery disease, cardiomyopathy, heart failure, valve diseases, arrhythmia) and in a stable condition
* No physical and/or mental condition that would prevent completing the scales
* Literate in Turkish

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria will be excluded.
* Participants who are found to have incomplete responses to the scale questions after being included in the study, as well as those who choose to withdraw from the study voluntarily, will be removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals with stable CVD who are outpatients at the cardiology clinics of Kırıkkale University Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Depression | Baseline
  The primary outcome measure in the study is depression, as determined by the Cardiac Depression Scale (CDS), while other scales and participant demographic data will be considered as independent variables. CDS scores range from 26 to 182, with higher scores indicating more severe depressive symptoms. A score of 95 or higher on the CDS can detect major depression in individuals with CVD with 85% specificity and 97% sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University Faculty of Medicine, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the study period will be shared.
Supporting Information: CSR

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Thombs BD, de Jonge P, Coyne JC, Whooley MA, Frasure-Smith N, Mitchell AJ, Zuidersma M, Eze-Nliam C, Lima BB, Smith CG, Soderlund K, Ziegelstein RC. Depression screening and patient outcomes in cardiovascular care: a systematic review. JAMA. 2008 Nov 12;300(18):2161-71. doi: 10.1001/jama.2008.667. PMID 19001627
- [Background] Hare DL, Selvadurai LP, Wang JQ, Yau HH, Stone MJ, Raman B, Wu N, Shi WY, Toukhsati SR. Psychometric assessment of the Cardiac Depression Scale Short Form in cardiac outpatients. Eur J Cardiovasc Nurs. 2017 Mar;16(3):249-255. doi: 10.1177/1474515116652759. Epub 2016 Jul 7. PMID 27231395
- [Background] Shi WY, Stewart AG, Hare DL. Major depression in cardiac patients is accurately assessed using the cardiac depression scale. Psychother Psychosom. 2010;79(6):391-2. doi: 10.1159/000320897. Epub 2010 Sep 9. No abstract available. PMID 20829653
- [Background] Wise FM, Harris DW, Carter LM. Validation of the Cardiac Depression Scale in a cardiac rehabilitation population. J Psychosom Res. 2006 Feb;60(2):177-83. doi: 10.1016/j.jpsychores.2005.07.019. PMID 16439271
- [Background] Kiropoulos LA, Meredith I, Tonkin A, Clarke D, Antonis P, Plunkett J. Psychometric properties of the cardiac depression scale in patients with coronary heart disease. BMC Psychiatry. 2012 Dec 3;12:216. doi: 10.1186/1471-244X-12-216. PMID 23199307
- [Background] Gholizadeh L, Salamonson Y, Davidson PM, Parvan K, Frost SA, Chang S, Hare DL. Cross-cultural validation of the Cardiac Depression Scale in Iran. Br J Clin Psychol. 2010 Nov;49(Pt 4):517-28. doi: 10.1348/014466509X478709. Epub 2010 Mar 25. PMID 20346205
- [Background] Wang W, Thompson DR, Chair SY, Hare DL. A psychometric evaluation of a Chinese version of the Cardiac Depression Scale. J Psychosom Res. 2008 Aug;65(2):123-9. doi: 10.1016/j.jpsychores.2008.03.010. PMID 18655856
- [Background] Hare DL, Davis CR. Cardiac Depression Scale: validation of a new depression scale for cardiac patients. J Psychosom Res. 1996 Apr;40(4):379-86. doi: 10.1016/0022-3999(95)00612-5. PMID 8736418
- [Background] Sobolewska-Nowak J, Wachowska K, Nowak A, Orzechowska A, Szulc A, Plaza O, Galecki P. Exploring the Heart-Mind Connection: Unraveling the Shared Pathways between Depression and Cardiovascular Diseases. Biomedicines. 2023 Jul 5;11(7):1903. doi: 10.3390/biomedicines11071903. PMID 37509542
- [Background] Feng L, Li L, Liu W, Yang J, Wang Q, Shi L, Luo M. Prevalence of depression in myocardial infarction: A PRISMA-compliant meta-analysis. Medicine (Baltimore). 2019 Feb;98(8):e14596. doi: 10.1097/MD.0000000000014596. PMID 30813183
- [Background] Tully PJ, Baker RA, Knight JL. Anxiety and depression as risk factors for mortality after coronary artery bypass surgery. J Psychosom Res. 2008 Mar;64(3):285-90. doi: 10.1016/j.jpsychores.2007.09.007. PMID 18291243
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103